CLINICAL TRIAL: NCT07156370
Title: Study to Explore the Prevalence of Hypercortisolism in Patients With Type 2 Diabetes and Assess the Correlation Between Salivary Cortisol and Glucose Levels
Brief Title: Salivary Cortisol and Hypercortisolism in Type 2 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Principal Investigator, Professor, Chief Physician, Deputy Director, Shanghai 6th People's Hospital
Other Study IDs: 20250810
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hypercortisolism; Type 2 Diabetes (T2DM)
MeSH Terms: conditions — Cushing Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to explore the prevalence of hypercortisolism in a population with difficult to control type 2 diabetes despite receiving standard-of-care therapies. Additionally, the study will evaluate the correlation between salivary cortisol levels and glycemic control.

DETAILED DESCRIPTION:
Despite advanced treatments, many individuals with type 2 diabetes develop refractory disease, leading to poor glycemic control and a higher risk of complications. Hypercortisolism, which promotes hyperglycemia, may be a key contributing factor. A recent study found a 23.8% prevalence of hypercortisolism in patients with difficult to control type 2 diabetes, linking the condition to higher rates of cardiovascular disease. As stable salivary cortisol testing can effectively screen for this condition, this study has two aims. First, the study will evaluate the prevalence of hypercortisolism in patients with difficult to control type 2 diabetes and identify its associated risk factors. Second, the study will establish the correlation between salivary cortisol and glycemic levels in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80 years.
2. Meets the definition of difficult to control type 2 diabetes:

HbA1c level between 7.5% and 11.5%, AND Taking 3 or more anti-hyperglycemic drugs. OR Taking insulin and other anti-hyperglycemic drugs. OR Taking 2 or more anti-hyperglycemic drugs AND a.) the presence of 1 or more micro-vascular or macro-vascular complication (retinopathy, diabetic nephropathy and chronic kidney disease, diabetic neuropathy, atherosclerotic heart disease with diabetes); AND/OR b.) concomitant hypertension requiring 2 or more anti-hypertension medications.

Exclusion Criteria:

1. Patients with Type 1 diabetes, new-onset diabetes (<1 year duration), or other specific types of diabetes.
2. History of systemic glucocorticoid use within the last 3 months (inhaled or topical agents are not exclusionary).
3. Pregnant or lactating.
4. Presence of severe cardiac, hepatic, renal, or other major organ dysfunction.
5. History of acute diabetic complications, such as diabetic ketoacidosis or hyperosmolar hyperglycemic state, within the last 3 months.
6. Presence of diseases that significantly affect metabolism, such as malignancy or autoimmune disorders.
7. Inability to tolerate adhesive tape, severe skin conditions at the sensor placement site, or presence of a psychiatric illness or cognitive impairment that would interfere with study compliance.
8. A known diagnosis of Cushing's syndrome, or currently receiving treatment with any of the following: mifepristone, metyrapone, osilodrostat, ketoconazole, fluconazole, aminoglutethimide, etomidate, octreotide, larazotide, long-acting octreotide, or pasireotide.
9. Excessive alcohol consumption (defined as >14 units per week for males or >7 units per week for females).
10. Severe, untreated sleep apnea.
11. Night shift workers (defined as being awake between 11:00 PM and 7:00 AM).
12. Known allergy or severe reaction to dexamethasone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are enrolled from the Department of Endocrinology and Metabolism from Shanghai Sixth People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Hypercortisolism | Baseline (Screening)
  Prevalence (percentage) of patients with hypercortisolism defined by dexamethasone suppression test (DST) >1.8 μg/dL in patients with difficult to control type 2 diabetes, defined as HbA1c 7.5-11.5%, despite receiving standard-of-care therapies.

SECONDARY OUTCOMES:
Correlation between salivary cortisol and glycemic levels | One week
  Correlation between salivary cortisol and glycemic levels, including hemoglobin A1c, glycated ablumin, 1,5-anhydroglucitol and metrics derived from continuous glucose monitoring.
Levels of salivary cortisol | 8:00, 16:00, 23:00, and 8:00 on the following day
  Levels of salivary cortisol in patients with difficult to control type 2 diabetes measured by fluorescence immunoassay system

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No